CLINICAL TRIAL: NCT04551846
Title: The Influence of Polymeric Versus Oligomeric Enteral Feeding on Tolerance and Nutritional Status in Paediatric Intensive Care: Prospective Randomized Trial
Brief Title: The Influence of Polymeric Versus Oligomeric Enteral Feeding on Tolerance and Nutritional Status in Paediatric Intensive Care
Acronym: Polygomer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KDAR FN Brno 2020/10/2
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Enteral Feeding Intolerance
Keywords: Enteral feeding; Enteral nutrition; Paediatric patient; Oligomeric; Polymeric

STUDY DESIGN:
Intervention Model Description: Monocentric randomized controlled trial with 2 groups: interventional (oligomeric formula) and control (polymeric)
Who Masked: Participant
Masking Description: The patients and the legal guardians will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligomeric enteral feeding group (Experimental): Oligomeric enteral nutrition will be administered according to the study protocol
  Interventions: Dietary Supplement: Oligomeric enteral feeding
- Polymeric enteral feeding group (Active Comparator): Polymeric enteral nutrition will be administered according to the study protocol
  Interventions: Dietary Supplement: Polymeric enteral feeding

INTERVENTIONS:
Dietary Supplement: Oligomeric enteral feeding — Oligomeric enteral feeding will be administered to the PICU patients
  Other Names: Oligomeric enteral formula
  Arms: Oligomeric enteral feeding group
Dietary Supplement: Polymeric enteral feeding — Polymeric enteral feeding will be administered to the PICU patients
  Other Names: Polymeric enteral formula
  Arms: Polymeric enteral feeding group

SUMMARY:
Malnutrition is associated with negative impact on morbidity and mortality of critically ill patients. Therefore, in patients unable of peroral intake, the nutritional support is indicated. The preferred form of nutritional support is enteral, the more natural form, compared to parenteral. The enteral nutrition is cheaper and is associated with better outcomes and lower incidence of associated complications. The intolerance of enteral feeding is common in critically ill patients, and is associated with insufficient energy and protein intake, that could be linked with the complications such aspiration pneumonia. The optimization of enteral feeding tolerance is therefore one of the research priorities. Implementation of feeding protocols is associated with better tolerance. The enteral feeding could be administered as a oligomeric or polymeric formula. The are preliminary data from adult population pointing at better tolerance of oligomeric feeding formula.

DETAILED DESCRIPTION:
After Ethics Committee approval, all paediatric patients admitted to the paediatric intensive care unit (PICU) will underwent PICU screening. In case of eligible for inclusion in to the study, the baseline parameters a demographics will be evaluated together with the initial laboratory sampling after approval and singed the informed consent by the legal guardian of the patient. Patients will be randomized by the online randomizer to the oligomeric and polymeric enteral nutrition group.

Polymeric (control group): Patients indicated for at least 2 days of enteral nutrition by the gastric tube. The nutritional support will be initiated after initial haemodynamic stabilization (blood levels of lactate normalization, norepinephrine infusion <0,1 ug/kg/min) in the 48-hours interval from admission in form of bolus administration of polymeric formula 1ml/kg/dose. The gastric residual volume will be evaluated after 4 hours from bolus dose. In case of gastric residual volume lower than half of previously administered dose, the next dose will be doubled. In case of higher residual volume, the same amount will be administered with the metoclopramid (3 times per day). In case of persistent residual volume higher than half of initial dose in 12 hours, the erythromycin will be initiated for 3 days. The bolus enteral feeding will be administered at the predefined time 5/day (6:00, 10:00, 14:00, 18:00, 22:00). The las gastric decompression is planned ad 24:00. The aim is to reach energetic goal defined by Schofield equation.

Interventional (oligomeric group): Patients indicated for at least 2 days of enteral nutrition by the gastric tube. The nutritional support will be initiated after initial haemodynamic stabilization (blood levels of lactate normalization, norepinephrine infusion <0,1 ug/kg/min) in the 48-hours interval from admission in form of bolus administration of oligomeric formula 1ml/kg/dose. The gastric residual volume will be evaluated after 4 hours from bolus dose. In case of gastric residual volume lower than half of previously administered dose, the next dose will be doubled. In case of higher residual volume, the same amount will be administered with the metoclopramid (3 times per day). In case of persistent residual volume higher than half of initial dose in 12 hours, the erythromycin will be initiated for 3 days. The bolus enteral feeding will be administered at the predefined time 5/day (6:00, 10:00, 14:00, 18:00, 22:00). The las gastric decompression is planned ad 24:00. The aim is to reach energetic goal defined by Schofield equation.

ELIGIBILITY:
Inclusion Criteria:

* PICU patients indicated for nutritional support by enteral feeding (gastric or jejunal)

Exclusion Criteria:

* Enteral feeding contraindicated
* Persistent haemodynamic instability
* Informed consent not signed
* Acute pancreatitis
* Recent upper gastrointestinal surgery
* Gut perforation
* Ileus

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The amount of energy delivery at 7th day | on the 7th day after study inclusion
  The amount of delivered energy at 7th day according to the defined energy goal by derived from Schofield equation
The amount of protein delivery at 7th day | on the 7th day after study initiation
  The amount of protein delivered at 7th day according to the defined protein delivery goal by derived from Schofield equation

SECONDARY OUTCOMES:
The time needed to achieve the energy target | in 7 days after study initiation
  The time needed to achieve the energy target according to the Schofield equation
The time needed to achieve the protein target | in 7 days after study initiation
  The time needed to achieve the protein target according to the Schofield equation
The daily energy delivery | in 7 days after study initiation
  The daily amount of energy delivery
The daily gastric residual volume | in 7 days after study initiation
  The daily gastric residual volume
The mean gastric residual volume | in 7 days after study initiation
  The mean gastric residual volume
The time to first stool | in 7 days after study initiation
  The time to first stool from study initiation
The daily number of stool | in 7 days after study initiation
  The daily number of stool from study initiation
Nutritional parameters 1 - albumin | in 7 days after study initiation
  albumin plasmatic levels
Nutritional parameters 1 - prealbumin | in 7 days after study initiation
  prealbumin plasmatic levels

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof. MD., Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided